CLINICAL TRIAL: NCT02816047
Title: Indications for and Experience With the Wearable Cardioverter Defibrillator (WCD) - Austrian WCD Registry
Brief Title: Austrian Wearable Cardioverter Defibrillator Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Scherr Daniel, MD, Austrian Wearable Cardioverter Defibrillator Registry, Medical University of Graz
Other Study IDs: KardioScherr1
Record Dates: First submitted 2016-05-17; First posted 2016-06-28 (Estimated); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Heart Failure; Ventricular Dysfunction; Sudden Death; Sudden Cardiac Arrest; Ventricular Tachycardia; Ventricular Fibrillation
Keywords: wearable cardioverter defibrillator; LifeVest; sudden death; defibrillator
MeSH Terms: conditions — Heart Failure; Ventricular Dysfunction; Death, Sudden; Death, Sudden, Cardiac; Tachycardia, Ventricular; Ventricular Fibrillation | interventions — Registries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Registry — Observational study to describe WCD indications, event rates, inappropriate shock rates and follow up (including ICD rate, shock rate, morbidity and mortality) in all Austrian WCD patients

SUMMARY:
Background: The wearable cardioverter defibrillator (WCD) is an established treatment option for patients at high risk for ventricular tachycardia / ventricular fibrillation (VT/VF), either in whom this risk may only be temporarily present, or in patients at high risk for sudden cardiac death (SCD) or after VT/VF in whom an implantable cardioverter defibrillator (ICD is currently not possible for other reasons (infection, recent MI <40days, recent PCI/CABG < 3months etc.).

Methods: Comprehensive registry including all patients in Austria who received a WCD in 2010-2016.

DETAILED DESCRIPTION:
Observational study to describe WCD indications, event rates, inappropriate shock rates and follow up (including ICD rate, shock rate, morbidity and mortality) in all Austrian WCD patients

ELIGIBILITY:
Inclusion Criteria:

* patients, with a prescribed WCD according to guidelines in an austrian center

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Comprehensive registry including all patients in all Austrian centers who received a WCD in 2010-2016.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2014-11; Primary Completion 2021-12 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants treated with WCD-treated ventricular arrhythmias | during WCD wearing period; average of 1 year
  Number of participants treated with WCD-treated ventricular arrhythmias

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Scherr, Assoz. Prof., Principal Investigator — Medical University of Graz/ Division of Cardiology
Locations (1):
- Medical University of Graz/ Division of Cardiology, Graz, Austria

IPD SHARING:
Plan to Share IPD: Undecided
possible